CLINICAL TRIAL: NCT00175175
Title: Randomized Trial of Osteoporosis Intervention Strategies in Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other); Royal Alexandra Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHFMR #200100791
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Osteoporosis; Hip Fracture
Keywords: osteoporosis treatment; osteoporosis testing; hip fracture; quality improvement
MeSH Terms: conditions — Osteoporosis; Hip Fractures | interventions — Case Management

INTERVENTIONS:
Behavioral: Allied health professional-run osteoporosis service ("case-management")

SUMMARY:
Patients with hip fractures have suffered the most devastating consequence of osteoporosis; and yet, they are rarely if ever tested or treated for the condition, even though they remain at high risk of recurrent fracture.

We hypothesize that, compared with usual care, an allied health professional-run osteoporosis service (case management) will be able to increase testing and treatment of osteoporosis in patients at high risk of fracture.

DETAILED DESCRIPTION:
Patients with hip fractures have suffered the most devastating consequence of osteoporosis; and yet, they are rarely if ever tested or treated for the condition, even though they remain at high risk of recurrent fracture.

We hypothesize that, compared with usual care, an allied health professional-run osteoporosis service (case management) will be able to increase testing and treatment of osteoporosis in patients at high risk of fracture.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture patient > 50 years of age
* able to give consent (or proxy consent available)
* lives within health region
* no contraindications to bisphosphonate therapy

Exclusion Criteria:

* refuses to participate or consent
* dementia or delirium without a proxy consent available
* nursing home or longterm care
* pathologic fracture
* chronic glucocorticoid use
* already receiving prescription osteoporosis treatment (calcium and vitamin D do not preclude inclusion)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2002-03

PRIMARY OUTCOMES:
The proportion of patients taking bisphosphonate therapy within 6 months of hip fracture

SECONDARY OUTCOMES:
Proportion of patients taking prescription osteoporosis treatment at 6 months and 12 months
Proportion in receipt of a BMD test at 6 months and 12 months
Proportion still adherent to osteoporosis treatments at 6 months and 12 months
Proportion of patients with recurrent fractures at 6 months and 12 months
Cost effectiveness analyses

CONTACTS AND LOCATIONS:
Overall Officials: Sumit R Majumdar, MD, MPH, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospitals, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Morrish DW, Beaupre LA, Bell NR, Cinats JG, Hanley DA, Harley CH, Juby AG, Lier DA, Maksymowych WP, Majumdar SR. Facilitated bone mineral density testing versus hospital-based case management to improve osteoporosis treatment for hip fracture patients: additional results from a randomized trial. Arthritis Rheum. 2009 Feb 15;61(2):209-15. doi: 10.1002/art.24097. PMID 19177538
- [Derived] Majumdar SR, Lier DA, Beaupre LA, Hanley DA, Maksymowych WP, Juby AG, Bell NR, Morrish DW. Osteoporosis case manager for patients with hip fractures: results of a cost-effectiveness analysis conducted alongside a randomized trial. Arch Intern Med. 2009 Jan 12;169(1):25-31. doi: 10.1001/archinte.169.1.25. PMID 19139320
- [Derived] Majumdar SR, Beaupre LA, Harley CH, Hanley DA, Lier DA, Juby AG, Maksymowych WP, Cinats JG, Bell NR, Morrish DW. Use of a case manager to improve osteoporosis treatment after hip fracture: results of a randomized controlled trial. Arch Intern Med. 2007 Oct 22;167(19):2110-5. doi: 10.1001/archinte.167.19.2110. PMID 17954806